CLINICAL TRIAL: NCT02443610
Title: Hémorragies et Maladie Veineuse Thromboembolique du Post-partum : Epidémiologie, Etudes Des déterminants Cliniques et Biologiques
Brief Title: Haemorrhages and Thromboembolic Venous Disease of the Postpartum
Acronym: HEMOTHEPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: HEMOTHEPP ( RB 13.175)
Record Dates: First submitted 2015-05-05; First posted 2015-05-14 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Postpartum Hemorrhage; Venous Thromboembolism
Keywords: Postpartum Hemorrhage; Venous Thromboembolism; Pregnancy
MeSH Terms: conditions — Postpartum Hemorrhage; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the frequencey and the determinants of postpartum major complications (hemorrhage and thrombosis) up to 3 months after delivery in the maternity hospitals of Finistère (Bretagne - France)

DETAILED DESCRIPTION:
This is an analytical observational prospective multicenter cohort study , conducted on all the maternity hospitals in Finistère (Bretagne - France), with a biological collection.

This protocol allows to study all women at risk of PPH (Postpartum Hemorrhage) and postpartum venous thromboembolic disease, including maternity level 1-3 without case selection. The prospective nature of the study should provide a more detailed analysis of exposures in this particular population of women (risk factors related to the field, childbirth, the postpartum events ...).

The events of interest were PPH and venous thromboembolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Any woman giving birth and supported in one of Gynaecology Obstetrics services of a maternity Finistere.
* Women ≥ 16 at the time of the collection of non-opposition.
* For minor patients: understanding the patient and at least one parent.
* All births ≥ 15 weeks gestation.

Exclusion Criteria:

* Home Birth
* Expressed opposition to participation in this study.
* Childbirth under X.
* Parent (s) uninformed of the pregnancy of their child.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All women admitted for delivery in a maternity Finistère
Sampling Method: Non-Probability Sample
Enrollment: 20241 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Postpartum Hemorrhage | 2 days
  Volume of blood loss up to 48 hours after delivery and / or weight compresses collected at delivery, and / or diagnosis of the clinician
Symptomatic thromboembolic events | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: PAN PETESCH Brigitte, Principal Investigator — Unité d'Hémostase , Centre Régional de traitement de l'hémophilie et des maladies hémorragiques, CHRU de Brest (France)
Locations (6):
- France (6):
  - CH de Carhaix, Carhaix-Plouguer, Finistère
  - CHRU de Brest - Service de Gynécologie-obstétrique, Brest
  - Clinique Keraudren, Brest
  - CH de Landerneau, Landerneau
  - CH de Morlaix, Morlaix
  - CH Quimper, Quimper

REFERENCES:
- [Derived] Anouilh F, de Moreuil C, Tremouilhac C, Jacquot M, Salnelle G, Bellec V, Touffet N, Cornec C, Muller M, Dupre PF, Bellot C, Morcel K, Joliff DL, Drugmanne G, Gelebart E, Lucier S, Nowak E, Bihan L, Couturaud F, Tromeur C, Moigne EL, Pan-Petesch B. Family history of postpartum hemorrhage is a risk factor for postpartum hemorrhage after vaginal delivery: results from the French prospective multicenter Haemorrhages and Thromboembolic Venous Disease of the Postpartum cohort study. Am J Obstet Gynecol MFM. 2023 Sep;5(9):101062. doi: 10.1016/j.ajogmf.2023.101062. Epub 2023 Jun 19. PMID 37343695